CLINICAL TRIAL: NCT01467947
Title: Prospective Open-label Uncontrolled Multi-center Post-marketing Study to Assess Inhibitory Antibody Formation in Subjects With Congenital C1-INH Deficiency and Acute Hereditary Angioedema (HAE) Attacks Treated With Berinert® , a C1-esterase Inhibitor
Brief Title: Postmarketing Immunogenicity Study in HAE Subjects Treated With Berinert
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE1145_4001; 2010-024242-30 (EudraCT Number)
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2015-10

CONDITIONS: Hereditary Angioedema Types I and II
MeSH Terms: conditions — Hereditary Angioedema Types I and II | interventions — Complement C1 Inhibitor Protein; Water; Injections

ARMS (1):
- Berinert (Experimental)
  Interventions: Biological: Berinert, lyophilizate for IV application containing 500 IU C1-INH to be reconstituted with 10 mL water for injection

INTERVENTIONS:
Biological: Berinert, lyophilizate for IV application containing 500 IU C1-INH to be reconstituted with 10 mL water for injection — Individual treatment duration per subject is 9 months, irrespective of the number of treated attacks. Each attack that occurs in this time frame will be treated with 20 IU Berinert/kg body weight.

SUMMARY:
This is a prospective, international, multi-center, non-randomized, single arm, open-label, postmarketing study to investigate the formation of inhibitory anti-C1-INH antibodies in HAE subjects treated intravenously with Berinert. Individual treatment duration per subject is 9 months, irrespective of the number of treated attacks. All subjects will receive 20 IU Berinert/kg body weight per attack.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital C1-INH deficiency (HAE type I or II) and assessed by the investigator to likely require intravenous (IV) Berinert treatment during the study period.
* Male or female, ≥ 12 years of age at the time of signing informed consent.
* Written informed consent for study participation obtained before undergoing any study specific procedures.

Exclusion Criteria:

* Incurable malignancies in the last 6 months prior to study entry.
* Acquired angioedema due to C1-INH deficiency.
* All other types of angioedema not associated with C1-INH deficiency.
* Use of any C1-INH products other than Berinert within 30 days before the study, or planned use during the study.
* Immunization within 30 days prior to study entry.
* Autoimmune conditions requiring use of immunosuppressants during the study.
* Known or suspected hypersensitivity to C1-INH.
* Participation in any of the previous Berinert studies from which anti-C1-INH antibody results were submitted to the Food and Drug Administration.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Rojavin, Study Director — CSL Behring
Locations (4):
- MHAT "Tsaritsa Yoanna", Sofia, Bulgaria
- Semmelweis University, Budapest, Hungary
- Jagiellonian University, Krakow, Krakow, Poland
- Spitalul Clinic Judeţean Mureş,Secţia Clinică Medicină Internă,Compartimentul Alergologie şi Imunologie, Târgu-Mures, Mureș County, Romania

REFERENCES:
- [Result] Farkas H, Varga L, Moldovan D, Obtulowicz K, Shirov T, Machnig T, Feuersenger H, Edelman J, Williams-Herman D, Rojavin M. Assessment of inhibitory antibodies in patients with hereditary angioedema treated with plasma-derived C1 inhibitor. Ann Allergy Asthma Immunol. 2016 Nov;117(5):508-513. doi: 10.1016/j.anai.2016.08.025. Epub 2016 Oct 24. PMID 27788880

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 subjects were screened and enrolled in the study. 14 subjects did not experience an HAE attack before the study ended and so did not receive study treatment. 46 subjects started and completed the active treatment period of the study.
Groups:
- C1 Esterase Inhibitor: Subjects received 20 IU C1 Esterase Inhibitor (C1-INH)/kg body weight by slow intravenous infusion for each acute HAE attack requiring treatment during a 9-month period beginning after their first HAE attack while on study.
Period: Overall Study
Arm/Group | C1 Esterase Inhibitor
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- C1 Esterase Inhibitor: Subjects received 20 IU/kg C1 Esterase Inhibitor (C1-INH)/kg body weight by slow intravenous infusion for each acute HAE attack requiring treatment during a 9-month period beginning after their first HAE attack while on study.
Arm/Group | C1 Esterase Inhibitor
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 42
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (14.42)
Gender [Count of Participants; unit: Participants]
  Female | 32
  Male | 14
Region of Enrollment [Number; unit: participants]
  Romania | 15
  Hungary | 8
  Poland | 13
  Bulgaria | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Inhibitory Anti-C1-esterase-inhibitor Antibodies
Description: Subjects with no positive baseline result and at least one positive post-baseline result for inhibitory anti-C1-INH antibodies.
Time Frame: Baseline to approximately 9 months
Measure: Number; unit: subjects
Arm/Group | C1 Esterase Inhibitor
Number analyzed (Participants) | 46
subjects | 0

2. Secondary Outcome: Number of Subjects With Any (Inhibitory or Non-inhibitory) Anti-C1-esterase-inhibitor Antibodies
Description: Subjects with at least one positive result for inhibitory or non-inhibitory anti-C1-INH antibodies.
Time Frame: Baseline to approximately 9 months
Measure: Number; unit: Subjects
Arm/Group | C1 Esterase Inhibitor
Number analyzed (Participants) | 46
Subjects
  Antibodies detected on Day 1 (Baseline) | 9
  Antibodies detected post-baseline | 10
  Antibodies first detected at Month 3 | 2
  Antibodies first detected at Month 6 | 1
  Antibodies first detected at Month 9 | 1

ADVERSE EVENTS:
Time Frame: Baseline to approximately 9 months.
Arm/Group | C1 Esterase Inhibitor
Serious Adverse Events (participants affected / at risk) | 2/46
Other Adverse Events (participants affected / at risk) | 7/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C1 Esterase Inhibitor (N=46)
Hereditary angioedema (Congenital, familial and genetic disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C1 Esterase Inhibitor (N=46)
Hypotension (Vascular disorders) | 3 (3)
Headache (Nervous system disorders) | 6 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.